CLINICAL TRIAL: NCT06189027
Title: Epigenetic Regulation of Stress-related Genes in Relation to MDMA-Assisted Psychotherapy Treatment for Post-Traumatic Stress Disorder
Brief Title: Epigenetics and MDMA-Assisted Psychotherapy for PTSD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Principal Investigator, Rael Cahn, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UP-18-00343
Record Dates: First submitted 2018-10-30; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: PTSD
Keywords: MDMA; Psychotherapy; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDMA Assisted Psychotherapy (Active Comparator): A longitudinal course of psychotherapy with administration of MDMA on two occasions to assist with the psychotherapeutic process
  Interventions: Drug: MDMA; Behavioral: Psychotherapy
- Placebo Assisted Psychotherapy (Placebo Comparator): A longitudinal course of psychotherapy with administration of placebo on two occasions to assist with the psychotherapeutic process
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Drug: MDMA — Adjunctive administration of MDMA to assist psychotherapeutic process
  Arms: MDMA Assisted Psychotherapy
Behavioral: Psychotherapy — Psychotherapy aimed at assisting with PTSD symptom reduction

SUMMARY:
This is an add-on substudy to an already-approved clinical trial "A Multi-Site Phase 3 Study of MDMA-Assisted Psychotherapy for PTSD" (ClinicalTrials.gov Identifier: NCT03537014) which is to be a phase 3 clinical trial studying the efficacy of MDMA-Assisted Psychotherapy for Post Traumatic Stress Disorder. The parent study has been approved by Copernicus Group IRB and is being run by the MAPS Public Benefit Corporation, and is a randomized controlled trial comparing the clinical efficacy of MDMA-assisted psychotherapy to Placebo-assisted psychotherapy. The parent study will recruit participants with Post Traumatic Stress Disorder and involves 20 total study visits over the course of 18 weeks including 3 preparatory psychotherapy visits plus 3 separate treatment sessions involving psychotherapy plus the administration of MDMA vs. placebo and 3 follow up psychotherapy visits after each treatment session.

This substudy adds on the collection of saliva in a salivary DNA collection kit at baseline and after treatment to the parent study clinical trail so as to assess whether the MDMA-Assisted Psychotherapy exerts influence on the epigenetic regulation of stress-associated genes as assessed in the salivary epithelial and white blood cells of the research participants. We aim to further assess whether any such changes are correlated with improvements in PTSD symptoms.

DETAILED DESCRIPTION:
For a detailed description of the parent study see "A Multi-Site Phase 3 Study of MDMA-Assisted Psychotherapy for PTSD" (ClinicalTrials.gov Identifier: NCT03537014). The current substudy the site coordinators at participating sites in the multi-site phase 3 clinical trial will collect saliva from research participants in the parent study at the following time points:

1. Collect saliva prior to first MDMA (vs placebo) treatment session at the Baseline Visit 3 or Visit 4 for the Phase 3 parent study, prior to the first MDMA (vs placebo) treatment session.
2. Collect saliva following final MDMA (vs placebo) treatment session at Primary Outcome Visit 19 or Visit 20 in the Phase 3 parent study, approximately 18 weeks after the first MDMA (vs placebo) treatment session.

The collection of saliva will be accomplished using the Oragene DNA OG-500 salivary DNA kits (https://www.dnagenotek.com/ROW/products/collection-human/oragene-dna/500-series/OG-500.html).

The salivary samples take no more than 2-3 minutes to collect by passive drool into the salivary collection kit.

ELIGIBILITY:
Criteria

Inclusion Criteria:

(As per the parent Phase III Trial - "A Multi-Site Phase 3 Study of MDMA-Assisted Psychotherapy for PTSD" (ClinicalTrials.gov Identifier: NCT03537014)).

1. *Are at least 18 years old
2. *Are fluent in speaking an d reading the predominantly used or recognized language of the study site
3. *Are able to swallow pills
4. Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments, and non-drug psychotherapy sessions
5. Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached
6. Must agree to inform the investigators within 48 hours of any medical conditions and procedures
7. If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session. Adequate birth control methods include intrauterine device (IUD), injected or implanted hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e. condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom). Not of childbearing potential is defined as permanent sterilization, postmenopausal, or assigned male at birth.
8. Agree to the following lifestyle modifications (described in more detail in Section 4.3 Lifestyle Modifications): comply with requirements for fasting and refraining from certain medications prior to Experimental Sessions, not participate in any other interventional clinical trials during the duration of the study, remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures Medical History
9. *At Screening, meet DSM-5 criteria for current PTSD with a symptom duration of 6 months or longer
10. *At Screening, have at least severe PTSD symptoms in the last month based on PCL-5 total score of 50 or greater
11. *At Screening, may have well-controlled hypertension that has been successfully treated with anti-hypertensive medicines, if they pass additional screening to rule out underlying cardiovascular disease
12. *At Screening, may have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed
13. At Baseline, have at least severe PTSD per CAPS-5 and symptoms in the last month constituting a CAPS-5 Total Severity Score of 35 or greater.

Exclusion Criteria:

(As per the parent Phase III Trial - "A Multi-Site Phase 3 Study of MDMA-Assisted Psychotherapy for PTSD" (ClinicalTrials.gov Identifier: NCT03537014)).

Potential participants are ineligible to enroll in the protocol if they:

1. *Are not able to give adequate informed consent
2. Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders
3. Are likely, in the investigator's opinion and via observation during the Preparatory Period, to be re-exposed to their index trauma or other significant trauma, lack social support, or lack a stable living situation
4. Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session; or have previously participated in a MAPS-sponsored MDMA clinical trial
5. Have any current problem which, in the opinion of the investigator or Medical Monitor, might interfere with participation

   Psychiatric History
6. *Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment
7. *Have a history of or a current primary psychotic disorder, bipolar affective disorder type 1 assessed via MINI and confirmed via clinical interview or dissociative identity disorder assessed via DDIS and confirmed via clinical interview
8. *Have a current eating disorder with active purging assessed via MINI and confirmed via clinical interview
9. *Have current major depressive disorder with psychotic features assessed via MINI
10. *Meet DSM-5 criteria for active substance use disorder for any substance other than caffeine or nicotine assessed via combination of clinical judgment, MINI, AUDIT, DUDIT, drug test, and blood %carbohydrate-deficient transferrin (%CDT)
11. Have current Personality Disorders Cluster A (paranoid, schizoid, schizotypal), Cluster B (antisocial, borderline, histrionic, narcissistic), or Cluster C (avoidant, dependent, obsessive-compulsive) assessed via SCID-5-PD.
12. Any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS, and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled
13. Would present a serious risk to others as established through clinical interview and contact with treating psychiatrist
14. Require ongoing concomitant therapy with a psychiatric medication with exceptions described in Section 12.0: Concomitant Medications.

    Medical History
15. *Have evidence or history of significant (controlled or uncontrolled) hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, renal, gastrointestinal, immunocompromising, or neurological disease, including seizure disorder, or any other medical disorder judged by the investigator to significantly increase the risk of MDMA administration (participants with hypothyroidism who are on adequate and stable thyroid replacement will not be excluded). Note: if participants present with a history of glaucoma, enrollment would be allowed only with the approval of their ophthalmologist
16. *Have uncontrolled hypertension using the standard criteria of the American Heart Association (values of 140/90 milligrams of Mercury [mmHg] or higher assessed on three separate occasions)
17. *Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] corrected by Bazett's formula)
18. *Have a history of additional risk factors for Torsade de pointes ( e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
19. *Require use of concomitant medications that prolong the QT/QTc interval during Experimental Sessions. Refer to Section 12.0 Concomitant Medications.
20. *Have symptomatic liver disease
21. *Have history of hyponatremia or hyperthermia
22. *Weigh less than 48 kilograms (kg)
23. Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Epigenetic regulation of target genes | 4 months
  Quantify changes in methylation of glucocorticoid receptor NR3C1, the associated gene FKBP5, and Brain Derived Neurotrophic Factor (BDNF) as compared to placebo, in participants with PTSD.
Correlation between PTSD Symptoms and Epigenetic Changes | 4 months
  Correlations between changes in PTSD symptoms and methylation changes in target genes

CONTACTS AND LOCATIONS:
Overall Officials: Rael Cahn, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- Univeristy of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to information on how to enroll in the parent Phase III Trial — https://maps.org/research/mdma/ptsd/phase3

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT06189027/Prot_SAP_000.pdf